CLINICAL TRIAL: NCT05292378
Title: Carbon Dioxide (CO2): A Pilot Study of a Hypothesized Mechanism to Explain Cognitive Impairment
Brief Title: Carbon Dioxide (CO2) and Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Howard M. Kipen, MD, MPH, Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro2021001570
Record Dates: First submitted 2022-01-24; First posted 2022-03-23 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: Carbon Dioxide; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High CO2 Exposure first, then low CO2 exposure second. (Experimental): At the first study visit the subject is exposed to 2500 ppm CO2 for 2.5 hours and at the second study visit the subject is exposed to 600 ppm CO2 for 2.5 hours.
  Interventions: Other: 2500 ppm Carbon Dioxide; Other: 600 ppm Carbon Dioxide
- Low CO2 Exposure first, then high CO2 exposure second. (Sham Comparator): At the first study visit the subject is exposed to 600 ppm CO2 for 2.5 hours and at the second study visit the subject is exposed to 2500 ppm CO2 for 2.5 hours.
  Interventions: Other: 2500 ppm Carbon Dioxide; Other: 600 ppm Carbon Dioxide

INTERVENTIONS:
Other: 2500 ppm Carbon Dioxide — 2.5 hour exposure to 2500 ppm carbon dioxide
Other: 600 ppm Carbon Dioxide — 2.5 hour exposure to 600 ppm carbon dioxide

SUMMARY:
The purpose of the study is to better understand the biological mechanisms of carbon dioxide (CO2)-induced cognitive impairments.

DETAILED DESCRIPTION:
Participants will complete 2 study visits. Each study visit will consist of a 2.5-hour exposure session. Concentrations of CO2 during the exposure session will be either 600 ppm (control) or 2500 ppm (exposure). The order of the exposure sessions will be randomized and the exposure sessions will be at least one week apart. Up to two participants will take part in each exposure session.

During each exposure a neurobehavioral assessment (Strategic Management Simulations or SMS) will be administered. Venous blood (30 mL) will be collected from subjects immediately before entering the chamber and immediately after the exposure. A subset of subjects (n=12) will also undergo a 60-minute fMRI scan. Another subset of subjects (up to 10) will not complete the SMS during the exposures but will undergo computer-assisted intravital microscopy (CAIM) to exam the conjunctival microvasculature before and after the exposure.

ELIGIBILITY:
Inclusion Criteria:

* History of COVID-19 vaccination
* Weigh at least 110 pounds

Exclusion Criteria:

* Colorblindness
* Inability to hear verbal instructions
* Cardiovascular disease, including a history of stroke
* Diabetes requiring the use of insulin
* Pregnancy
* Current asthma (an asthma attack within the past five years)
* Medications for or history of anxiety disorder diagnosis or panic attacks
* Medications which may affect cognition such as beta-blockers and CNS depressants

Temporary Exclusion Criteria

* Respiratory symptoms in the previous four weeks
* Use of sedating cold/allergy medications in the previous week
* Use of marijuana in the previous week
* Consumption of alcohol in the previous 24 hours

Additional Exclusion Criteria for Subjects undergoing the fMRI scan:

* History of head trauma or neurosurgery or neurological disorder
* Ferrous metal implanted in or on the body, electrical devices such as a pacemaker, nonremovable ferrous jewelry
* Surgical pins or plates above the neck
* History of eye injury involving metallic materials, shavings in eyes, or welding without a face mask
* Lead or iron tatoos
* Claustrophobia
* Back problems that would prevent the subject from laying still comfortably for up to 90 minutes

Additional Exclusion Criteria for Subjects undergoing CAIM

* Current or recent contact lens use

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Change in PMN (polymorphonuclear leukocyte) activation from pre-exposure to post-exposure | Immediately before and immediately after each exposure
  Using blood samples collected pre- and post-exposure, PMN activation will be assessed by measurement of oxidative burst (oxygen consumption rate), glycolytic function (extracellular acidification rate) and caspase-1 activity (assessed by fluorometric assay).

CONTACTS AND LOCATIONS:
Overall Officials: Howard Kipen, MD, Principal Investigator — Professor
Locations (1):
- Rutgers - EOHSI, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

DOCUMENTS (1):
  • Informed Consent Form (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT05292378/ICF_000.pdf